CLINICAL TRIAL: NCT06052358
Title: Left Atrial Appendage Closure With WATCHMAN FLX Device in Recurrent Gastrointestinal Bleeding: The GI-FLX Registry
Status: Terminated | Type: Observational
Why Stopped: The study has been closed by the Sponsor.
Sponsor: Kansas City Heart Rhythm Research Foundation (Other)
Collaborators: Kansas City Heart Rhythm Institute, Overland Park, Kansas (Unknown); Texas Cardiac Arrythmia Institute, Austin, Texas (Unknown); Los Robles Health System, Los Robles, California (Unknown); Centennial Medical Center, Nashville, Tennessee (Unknown)
Responsible Party: Sponsor
Other Study IDs: KCHRRF_GI FLX_0022
Record Dates: First submitted 2023-09-18; First posted 2023-09-25 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Atrial Fibrillation; GI Bleeding
MeSH Terms: conditions — Atrial Fibrillation; Gastrointestinal Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (2):
- Patients with a history of AF and GI bleeding who will undergo LAAC: This is group of patients who will undergo LAAC with Watchman FLX device and have a history of AF and GI bleed.
  Interventions: Device: LAAC with Watchman FLX device
- Patients with a history of AF and GI bleeding without LAAC: This is a historical cohort of patients with AF and recurrent GI bleeding without LAAC.

INTERVENTIONS:
Device: LAAC with Watchman FLX device — LAAC with Watchman FLX device
  Groups: Patients with a history of AF and GI bleeding who will undergo LAAC

SUMMARY:
The GI-FLX Registry is intended to create a registry of patients with a history of Atrial Fibrillation (AF) and Gastrointestinal (GI) bleed who will receive Left Atrial Appendage Closure (LAAC) with WATCHMAN FLX device and compare to patients with AF and GI bleed who do not have LAAC. The GI-FLX Registry will be a multi-center, non-randomized registry. Approximately 250 prospective patients will be enrolled at all 4 sites. Historical cohort of 250 patients after propensity score matching with WATCHMAN-FLX arm will be included in the final analysis.

DETAILED DESCRIPTION:
A large gap in the literature exists as no prior study has evaluated the outcomes of those with prior GI bleeding undergoing LAAC. Furthermore, patients with prior GI bleed may be on no or minimal antithrombotic therapy prior to LAAC and subsequently require escalation of antithrombotic therapy following LAAC. Long-term outcomes including bleeding events will be most relevant and informative to this potentially high-risk subgroup. Therefore, this is an attempt to create a prospective registry describing outcomes of patients with AF and prior GI bleed undergoing LAAC to provide insight into safety and efficacy and will also compare to a historical cohort of patients with AF and GI bleed without LAAC.

ELIGIBILITY:
Inclusion Criteria:

* All male and female patients who are > 18 years of age
* Have Atrial Fibrillation
* Have CHADS2VASc > 2
* Have history of GI bleeding OR hospital admission that required blood transfusion OR emergency room visit requiring stopping of OAC OR outpatient 2 gm of Hgb drop from baseline, with or without evidence of upper or lower GI bleeding and requiring endoscopic procedure with holding of OAC.
* Ability to understand study procedures and to comply with them for the entire length of the study.

Exclusion Criteria:

* Inability or unwillingness of individual to give written informed consent.
* Other indications for OAC like deep vein thrombosis (DVT) or Pulmonary embolism (PE) or mechanical heart valve.
* Patient who is pregnant will be excluded (Pregnancy will be excluded by checking urine beta-HCG).
* Patient not following up with our practice / clinic after the procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Approximately 250 patients who will undergo LAAC with Watchman FLX device and have a history of AF and GI bleed will be enrolled. This group will be compared to a historical cohort group of 250 patients with AF and recurrent gastrointestinal bleeding without LAAC.
Sampling Method: Non-Probability Sample
Enrollment: 73 (Actual)
Dates: Start 2023-08-23 (Actual); Primary Completion 2025-06-11 (Actual); Study Completion 2025-06-11 (Actual)

PRIMARY OUTCOMES:
Number of participants with Primary systemic thromboembolism (STE)/stroke, Recurrent bleeding after initial period of oral anticoagulant (OAC) requiring blood transfusion or hospitalization and Hemorrhagic stroke | 12 Months
  Baseline characteristics of participants such as Primary systemic thromboembolism (STE)/stroke, Recurrent bleeding after initial period of oral anticoagulant (OAC) requiring blood transfusion or hospitalization and Hemorrhagic stroke will be evaluated

SECONDARY OUTCOMES:
Number of participants with complications such as Peri-device leaks (PDL), Device related thrombosis (DRT), Minor bleeding episodes leading to hospital visit but no transfusion, Incidence of hospitalization and Mortality | 45 Days, 6 Months and 12 Months
  Number of participants with complications such as Peri-device leaks (PDL), Device related thrombosis (DRT), Minor bleeding episodes leading to hospital visit but no transfusion, Incidence of hospitalization and Mortality will be evaluated.
Number of days or hours of Hospital stay | 45 Days, 6 Months and 12 Months
  If any participants are hospitalized, their Hospital length of stay will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Dhanunjaya Lakkireddy, MD, Principal Investigator — Kansas City Heart Rhythm Institute
Locations (4):
- United States (4):
  - Kansas City Heart Rhythm Institute - Roe Clinic, Overland Park, Kansas
  - Overland Park Regional Medical Center, Overland Park, Kansas
  - Research Medical Center Clinic, Kansas City, Missouri
  - Research Medical Center, Kansas City, Missouri

REFERENCES:
- [Background] Decision Memo for Percutaneous Left Atrial Appendage (LAA) Closure Therapy (CAG- 00445N). Washington, DC: Centers for Medicare & Medicaid Services, 2016. In.
- [Background] Holmes DR, Reddy VY, Turi ZG, Doshi SK, Sievert H, Buchbinder M, Mullin CM, Sick P; PROTECT AF Investigators. Percutaneous closure of the left atrial appendage versus warfarin therapy for prevention of stroke in patients with atrial fibrillation: a randomised non-inferiority trial. Lancet. 2009 Aug 15;374(9689):534-42. doi: 10.1016/S0140-6736(09)61343-X. PMID 19683639
- [Background] Holmes DR Jr, Kar S, Price MJ, Whisenant B, Sievert H, Doshi SK, Huber K, Reddy VY. Prospective randomized evaluation of the Watchman Left Atrial Appendage Closure device in patients with atrial fibrillation versus long-term warfarin therapy: the PREVAIL trial. J Am Coll Cardiol. 2014 Jul 8;64(1):1-12. doi: 10.1016/j.jacc.2014.04.029. PMID 24998121
- [Background] Darden D, Duong T, Du C, Munir MB, Han FT, Reeves R, Saw J, Zeitler EP, Al-Khatib SM, Russo AM, Minges KE, Curtis JP, Freeman JV, Hsu JC. Sex Differences in Procedural Outcomes Among Patients Undergoing Left Atrial Appendage Occlusion: Insights From the NCDR LAAO Registry. JAMA Cardiol. 2021 Nov 1;6(11):1275-1284. doi: 10.1001/jamacardio.2021.3021. PMID 34379072